CLINICAL TRIAL: NCT06932510
Title: EFFECTS OF INFLATTABLE CERVICAL TRACTION COLLAR AS COMPARED TO MANUAL TRACION IN THE MANAGEMENT OF CERVICAL RADICULOPATHY
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Muhammad Osama, Assistant Professor, Foundation University Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/5
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor are blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Traction (Active Comparator): "Manual Traction Group" will be given Manual Traction with facet joint and Upper Extremity Neural Mobilization with Hot Pack and electrotherapy for 20 minutes.
  Interventions: Procedure: Manual Traction
- Cervical Traction Collar (Experimental): "Cervical Traction Collar" will be given Manual Traction with facet joint and Upper Extremity Neural Mobilization with Hot Pack and electrotherapy for 20 minutes.
  Interventions: Device: Cervical Traction Collar

INTERVENTIONS:
Procedure: Manual Traction — Manual cervical traction will be administered by a trained physical therapist.
  Arms: Manual Traction
Device: Cervical Traction Collar — Cervical traction will be administered via Cervical Traction Collar.
  Arms: Cervical Traction Collar

SUMMARY:
This study is a randomized control trial and the purpose of this study is to determine the effects of inflatable cervical traction collar as compared to manual traction in the management of cervical radiculopathy.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of inflatable cervical traction collar as compared to manual traction in the management of cervical radiculopathy on

1. Pain
2. Functional Disability
3. Range of motion Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Recruited participants will be allocated to either of the groups through a sealed opaque envelope method.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 19-44 years Neck pain >4 and <8 on NPRS NDI scoring <24(moderate disability) Positive Spurling test Positive Distraction Test Active and passive ROM limited/painful towards the side of pain Radiating Symptoms Numbness/paresthesia radiating to upper limb Both genders Positive - Upper Limb Neural Tension Tests (ULNTT) will be included. -

Exclusion Criteria:

Patients having Bilateral radiating sign and symptoms Cervical myelopathy Cervical syringomyelia Rheumatoid arthritis Thoracic outlet syndrome Brachial plexopathy Cervical Rib Vertebrobasilar insufficiency Recent history of fracture, surgery, trauma or whiplash Positive alar ligament stress test Positive sharp purser stress test Cervical instability Cancer, tumor or sudden weight loss.

-

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Neck Pain | 2 weeks
  Neck pain will be measured using Visual Analogue Scale, which has scoring from 0 to 100 mm, and a higher score represents greater pain and a lower score represents less pain.
Neck Disability Index | 2 weeks
  It consists of 10 items, each scored on a scale of 0-5, with 0 indicating no pain or limitations and 5 indicating the worst imaginable pain or limitation. The total score ranges from 0-50, with higher score indicating greater disability. The score can also be expressed in terms of percentage.
Cervical Range of Motion | 2 weeks
  Cervical range of motion will be measured using a Goniometer. A higher score represents greater range of motion, and lower score represents decreased or lesser range of morion of cervical spine.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Iqbal, DPT, Principal Investigator — Foundation University Islamabad; Muhammad Osama, PhD, Study Director — Foundation University Islamabad
Locations (1):
- Foundation University College of Physical Therapy, Foundation University Islamabad., Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No